CLINICAL TRIAL: NCT06275516
Title: A Single-blind Randomized Controlled Trial of Multisensory Stimulation Virtual Reality to Improve Motor and Cognitive Function in Stroke Patients
Brief Title: Safety and Efficacy of Multisensory Stimulation Virtual Reality for Stroke Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dingqun Bai, First Affiliated Hospital of Chongqing Medical University, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-208
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR+treadmill training group (Experimental): Multi-sensory stimulation immersive VR+ treadmill training with suitable for training intensity. 20 minutes a day for 30 days, a total of 600 minutes (training frequency is adjusted according to the patient's own conditions).
  Interventions: Device: multi-sensory stimulation immersive VR+ treadmill training
- treadmill training group (Active Comparator): Only treadmill training similarly with suitable for training intensity in the control group. 20 minutes a day for 30 days, a total of 600 minutes (training frequency is adjusted according to the patient's own conditions).
  Interventions: Device: treadmill training

INTERVENTIONS:
Device: multi-sensory stimulation immersive VR+ treadmill training — Treadmill training with multi-sensory stimulation immersive VR in VR+treadmill training group
  Arms: VR+treadmill training group
Device: treadmill training — Only treadmill training in treadmill training group
  Arms: treadmill training group

SUMMARY:
This was a single-blind randomized controlled trial of multisensory stimulation virtual reality to improve motor and cognitive dysfunction in stroke patients.

DETAILED DESCRIPTION:
This was single-blind randomized controlled intervention study. Each stroke subject underwent screening period, baseline assessment period, intervention period, endpoint assessment period.

The screening period include the verification of inclusion/exclusion criteria and the acquisition of informed consent.

Baseline and endpoint assessment period include motor function related scales were evaluated (muscle strength, muscle tone, Fugl-Meyer scale, Berg balance scale); cognitive function related scale assessment [Brief Mental State Examination Scale (MMSE), Montreal Cognitive Assessment (MoCA), drawing clock test, Shape connection test A.B, standardized digital modal experiment, auditory word Learning Test], emotional correlation scale assessment (Hamilton Depression Scale, Hamilton Anxiety Scale), and activity of daily living scale ADL scale. Meanwhile, quantitative evaluation of motor function three-dimensional gait detection and assessment of brain functional activation (fNIRs tests and fMRI) were synchronously completed.

The intervention period included multi-sensory stimulation immersive VR+ treadmill training with suitable for training intensity in the experimental group and only treadmill training similarly with suitable for training intensity in the control group. 20 minutes a day for 30 days, a total of 600 minutes (training frequency is adjusted according to the patient's own conditions).

Preliminary validation of effectiveness assessment includes Fugl-Meyer scale, Berg balance scale, and three-dimensional gait detection. Preliminary validation of the safety assessment includes fall and dizzy incidents.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stroke by neuroimaging (CT or MRI) assessment
2. 18-85 years old
3. Be able to walk with minor assistance
4. Can tolerate the rehabilitation training of this experiment
5. First stroke
6. Be able to follow instructions to complete the test
7. Patients who signed informed consent

Exclusion Criteria:

1. The test could not be tolerated due to organic disease
2. There is a serious mental illness resulting in inability to cooperate with or tolerate this test
3. is participating in another clinical trial involving an investigational drug or physical therapy
4. Patients who have not signed informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer scale | 30 days (Adjust according to the actual situation of patients)
  Motor function assessment
Berg balance scale | 30 days (Adjust according to the actual situation of patients)
  Balance function evaluation
three-dimensional gait detection | 30 days (Adjust according to the actual situation of patients)
  Quantitative motor function assessment
Fall incidents | 30 days (Adjust according to the actual situation of patients)
  Safety assessment
Dizzy incidents | 30 days (Adjust according to the actual situation of patients)
  Safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Dingqun Bai, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, First Branch, Chongqing, Chongqing Municipality, China